CLINICAL TRIAL: NCT01425398
Title: A Randomized, Double-Blinded, Placebo-Controlled Study Evaluating the Effect of Rosuvastatin on Inflammation in Patients Undergoing Isolated Cardiac Valve Surgery
Brief Title: A Trial to Evaluate the Effect of Rosuvastatin on Inflammation in Patients Undergoing Isolated Cardiac Valve Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jacques Genest, Co-Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: statins_inflammation_CVsurgery
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Valvular Cardiac Surgery
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin 40 mg PO qd x 5 days before surgery and then from post-op day 0 to 5.
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Placebo 1 tab qd x 5d before operation and then from post-op day 0 to 5
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 40 mg PO qd x 5 days before surgery and then from post-op day 0 to 5.
  Other Names: Rosuvastatin 40 mg/day
  Arms: Rosuvastatin
Drug: Placebo — Placebo 1 tab qd x 5d before operation and then from post-op day 0 to 5.
  Arms: Placebo

SUMMARY:
High-dose statin therapy around the time of surgery, decreases inflammation in patients undergoing cardiac valve surgery, and thereby improves clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple valve repairs or replacements without coronary artery bypass grafting
* Bentall procedure, but no other aortic procedures
* With or without accompanying MAZE procedure (surgical treatment for atrial fibrillation)

Exclusion Criteria:

* Age under 18 years old
* Urgent or emergency surgery
* Unable to provide consent
* Presently on statin therapy or exposure to statins within a month of surgery
* Chronic anti-inflammatory use, including steroids and NSAID's (nonsteroidal anti-inflammatory drugs) (not to be used during the treatment period)
* Known hypersensitivity to rosuvastatin
* Active liver disease Indicated by AST/ALT higher than 3 times the upper limit of normal
* Pregnant or nursing women
* On drugs with interactions (Cyclosporine, gemfibrozil, lopinavir/ritonavir or atazanavir/ritonavir, niacin) Severe renal impairment not on dialysis
* Creatinine clearance < 30 ml/min/1.73 m2
* Known myopathy and inflammatory diasthesis (such as systemic lupus erythromatosus, rheumatoid arthritis, and inflammatory bowel disease)
* Human Immunodeficiency Virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Improved Inflammatory Markers | Within 5 days post-op and at 3 months
  Significant (p<0.05) improvement of measured inflammatory markers

SECONDARY OUTCOMES:
Mortality | Within 3 months
  Significant (p<0.05) reduction of mortality in rosuvastatin arm versus placebo
Stroke | Within 3 months
  Significant (p<0.05) reduction of stroke events in rosuvastatin arm versus placebo
Myocardial Infarction | Within 3 months
  Significant (p<0.05) reduction of MI events in rosuvastatin arm versus
ICU length of stay | 3 months
  Significant reduction (p<0.05) of length of stay in rosuvastatin arm versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Genest, MD, Principal Investigator — RI-MUHC
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada